CLINICAL TRIAL: NCT06691087
Title: ÉTude de la pERception soNorE de Personnes maLentendantes équipées d'Aides Auditives
Brief Title: Sound Perception Study of Hearing-impaired People With Hearing Aids
Acronym: ETERNEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de l'Audition (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-040; 2024-A01112-45 (Other: ID-RCB)
Record Dates: First submitted 2024-10-14; First posted 2024-11-15 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Auditory Perception
MeSH Terms: interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Hearing participants (Active Comparator)
  Interventions: Behavioral: Influence of the parameters of the sound timbre on the perception of a sound; Behavioral: Complex sound scene comprehension test
- Hearing-impaired with hearing aids (Experimental)
  Interventions: Behavioral: Influence of the parameters of the sound timbre on the perception of a sound; Behavioral: Complex sound scene comprehension test; Behavioral: Complex sound scene comprehension test with hearing aids

INTERVENTIONS:
Behavioral: Influence of the parameters of the sound timbre on the perception of a sound — The experiment consists of evaluating the sound level of n complex stimuli, then equalising them in loudness, in order to measure a loudness curve in function of timbre descriptors.
  The stimuli will then be listened to again in pairs. The task is there to compare the stimuli using a VAS to indicate how different the two sounds are.
Behavioral: Complex sound scene comprehension test — The experiment consists in identifying the parameters of the sound timbre that most disturb the understanding of complex sound scenes, by asking the participants to identify sounds whose timbre has been modified.
Behavioral: Complex sound scene comprehension test with hearing aids — The experiment will be identical to intervention 2. This time, the modification of the stimulus timbres will focus on the most problematic dimensional modifications, i.e. those where the difference between normal-hearing and hearing-impaired listeners is greatest. We will then modify the signal processing parameters of the hearing aid simulator (for example, the size of the averaging window or the gain balance of the filters), to observe their impact on the salience of certain stimuli.
  Arms: Hearing-impaired with hearing aids

SUMMARY:
The aim of the ETERNEL project will be to study the influence of the perception of a single sound timbre on the understanding of a complex sound scene in hearing-impaired people with hearing aids. This will be done by quantifying the inability to manage a complex sound scene as a function of the timbre of the sounds making it up. The more a sound interferes with understanding the complex sound scene, the more salient that sound is considered to be. In this way, the investigators can determine which timbre dimensions make sounds particularly salient for the hearing impaired.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age between 60 and 75
* Native French speaker
* Have given their consent to take part in the study.
* Declare that they have an active social life or hobbies that stimulate their cognitive abilities
* Have a MOCA score above 26
* No tympano-ossicular dysfunction.
* Voice in noise audiometry results showing normal results.

For participants with impaired hearing :

* Pure tone audiometry showing audiograms of type N3 or N4 and symmetrical between the two ears.
* Report having experienced problems with abnormally prominent sound.

For participants with normal hearing:

- Pure tone audiometry showing audiograms with losses of less than 30 dBHl.

Exclusion Criteria:

* Be under guardianship or curatorship,
* Be deprived of liberty by judicial or administrative decision, or be under legal protection.
* Bear the consequences of an ear infection and/or have a history of an ENT disease that permanently affects hearing or balance (vestibular schwannoma, Ménière's disease, sudden or fluctuating deafness, congenital hypoacusis).

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of correct answers in melody comparison tasks in the hearing-impaired group compared with the normal-hearing group, | 3-hours

SECONDARY OUTCOMES:
Characterisation of the dissimilarity between pairs of stimuli measured by a continuous perceptual scale | 3-hours
  Continuous perceptual scale ranging from very dissimilar to very similar
Evaluation of the perceived loudness level of a set of stimuli, measured using scales of magnitude. | 3-hours
  11-point Likert scale
Comparison between the results of speech audiometry in noise, i.e number of words correctly repeated, with native settings versus settings minimising the discomfort of salient sounds for each participant with hearing loss. | up to 24 months
  the comparison will focus on the number of words correctly repeated on the 1st visit (with native settings) versus the last visit (with settings minimising the discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Avan, Principal Investigator — CERIAH

IPD SHARING:
Plan to Share IPD: No